CLINICAL TRIAL: NCT05889910
Title: Effectiveness of the Implementation of a Standardized Care Plan to Improve Fear of Falling and Incidence of Falls. FEARFALL_CARE Study
Brief Title: Effectiveness of the Implementation of a Standardized Care Plan to Improve Fear of Falling and Incidence of Falls
Acronym: FFC23
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Nuria Alcolea Ruiz, Enfermera Especialista en Atención Familiar y Comunitaria. Master Oficial de Investigación en Cuidados de Salud. Doctoranda en el Programa de Cuidados en Salud de la Universidad Complutense de Madrid., Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEARFALL_CARE
Record Dates: First submitted 2023-05-08; First posted 2023-06-05 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-11

CONDITIONS: Falls; Fear of Falling; Nursing
Keywords: Health Primary Care

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, multicenter, cluster-randomized clinical trial, 1:1 participant distribution ratio.
Who Masked: Outcomes Assessor
Masking Description: To avoid selection bias, professionals were blinded to group assignment at the time of patient recruitment.
  Once everyone had signed the informed consent, a cluster group was assigned to each of the 10 participating Health Centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention will consist of 5 initial sessions, plus a reinforcement session at 6 months. The sessions will last 2 hours and will preferably be distributed one day a week.
  To this end, nursing interventions will be included to improve the knowledge, skills and attitudes of the participants regarding the improvement of their functional capacity, the prevention of falls and their preventive measures, as well as the improvement in the management of anxiety and coping with the fear of falling and falls.
  The activities carried out during the intervention have been extracted from standardized nursing interventions through the Nursing Interventions Classification (NIC).
  The following interventions and activities will be addressed: 1665, 5612, 6490, 6486, 4700, 5820 and 5230.
  Interventions: Procedure: Health education workshop
- Control Group (Active Comparator): The control group intervention will be the usual clinical practice offered by the patient's nurse in the Primary Care setting during the duration of the study.
  The usual clinical practice is based on attention to the user's demands, as well as the performance of interventions that can influence falls and/or the fear of falling. These activities or interventions are based on the Services of the Standardized Service Portfolio of the Community of Madrid (Updated as of January 28, 2022) in which these patients are included due to age or as a consequence of their chronic pathology.
  Interventions: Procedure: Health education workshop

INTERVENTIONS:
Procedure: Health education workshop — The intervention will consist of 5 initial sessions, plus a reinforcement session at 6 months. The sessions will last 2 hours and will preferably be distributed one day a week.
  The objective of the intervention is to reduce the fear of falling and falls in people over 65 years of age who live in the community. To this end, nursing interventions will be included to improve the knowledge, skills and attitudes of the participants regarding the improvement of their functional capacity, the prevention of falls and their preventive measures, as well as the improvement in the management of anxiety and coping with the fear of falling and falls.
  The activities carried out during the intervention have been extracted from standardized nursing interventions through the Nursing Interventions Classification (NIC).
  The following interventions and activities will be addressed: 1665, 5612, 6490, 6486, 4700, 5820 and 5230.

SUMMARY:
The objective of this clinical trial is to evaluate the effectiveness of the implementation of a standardized care plan to reduce the fear of falling in people over 65 years of age with fear of falling who live in the community.

The main questions it aims to answer are:

* Is it possible to reduce the fear of falling in patients over 65 years of age through an educational intervention in primary care?
* Is it possible to reduce falls in patients older than 65 years through an educational intervention in primary care?

Half of the participants will receive an educational intervention consisting of 6 two-hour sessions at the Health Center. The comparison group will follow the usual clinical practice recommended by the Primary Care Assistance Management of the Community of Madrid. It is intended to observe if there are differences in the fear of falling and falls in both groups.

DETAILED DESCRIPTION:
General objective: To evaluate the effectiveness of the implementation of a standardized care plan to reduce the fear of falling in people over 65 years of age with fear of falling who live in the community.

Specific objectives:

* Determine the score of the short FES-I questionnaire in people over 65 years of age who have completed the care plan and in those who have followed usual clinical practice.
* Analyze the relationship between the sociodemographic variables of the patients and the clinical and functional variables with the score of the short FES-I questionnaire, both in the control and intervention groups.
* Analyze the relationship between the sociodemographic variables of the patients and the clinical and functional variables with the incidence of falls in both the control and intervention groups.
* Analyze the satisfaction of the application of the proposed standardized care plan.
* Analyze the safety of the application of the proposed standardized care plan.
* Analyze the effect of the intervention (measured through the mean difference in the short FES-I questionnaire) on the functional variables, the emotional state (anxiety and depression, measured through the Generalized Anxiety Disorder-7 (GAD- 7) and Patient Health Questionnaire-8 (PHQ-8)), self-care capacity (through the Self-Care Agency Capacity-Reduced scale) and perception of health.
* Characterize (by age, sex, functional status, clinical and emotional situation) the patients who suffered falls.
* Evaluate the feasibility and acceptability by patients and professionals of carrying out a Randomized Clinical Trial (RCT) to reduce the fear of falling and the incidence of falls by carrying out a standardized care plan that combines physical exercise and cognitive therapy. behavioral.

ELIGIBILITY:
Inclusion Criteria:

* People over 65 years of age on the start date of the study.
* People who are independent for the basic activities of daily living (ABVD) or who have mild functional dependence (Barthel Index score ≥ 60 and Short Physical Performance Battery (SPPB) ≥ 4),
* independent for ambulation (they walk 45m without help or with a cane),
* without cognitive impairment (Mini-Mental State Examination ((MMSE) ≥ 24).
* and with fear of falling (Short FES-I ≥ 11).

Exclusion Criteria:

* People with the following medical diagnoses or health problems (coded according to the International Classification of Diseases (ICD - 10):

  - Diagnosis of mental, behavioral and neurodevelopmental disorders: delirium, dementia, amnestic disorders and other cognitive disorders (F05.0; F05.9; F00; F02.8; F03; F04; R41.3; F06.9). Mental disorders due to general medical condition, unclassified in other sections (F06.1; F07.0; F09). Schizophrenia and other psychotic disorders (F20; F22; F23; F24; F29).
  * Diagnosis of neurodegenerative diseases: Parkinson's disease (G20); Alzheimer's disease (G30); Multiple sclerosis (G35); Myasthenia gravis and other myoneuronal disorders (G70).
  * Diagnosis of blindness and low vision (H54).
  * Diagnosis of conductive and sensorineural hearing loss bilateral or uncorrected with a hearing aid (H90.0; H90.2; H90.5; H90.6; H90.8) and other types of hearing loss, (H83.3; H91) whenever they make it difficult for the participants to understand.
  * Diagnosis of acute ischemic heart diseases and cerebrovascular diseases in the last 1 year (I20-I24; I60-I63; I67; I68).
* Hospitalization during the recruitment period or forecast admissions scheduled during the study period.
* Institutionalized patients or with frequent changes of address.
* Refusal to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 163 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Short Falls Efficacy Scale-International adapted to Spanish. | One month post intervention.
  (FES-I) Range 7-28. 11 or more points: indicates fear of falling.
Short Falls Efficacy Scale-International adapted to Spanish. | Six months post intervention.
  (FES-I)Range 7-28. 11 or more points: indicates fear of falling.
Short Falls Efficacy Scale-International adapted to Spanish. | 12 months post intervention.
  (FES-I). Range 7-28. 11 or more points: indicates fear of falling.

SECONDARY OUTCOMES:
Number of participants with post-intervention Falls. | One month post-intervention.
  Post-intervention Falls (yes or no)
Number of participants with post-intervention Falls. | Six months post intervention.
  Post-intervention Falls (yes or no)
Number of participants with post-intervention Falls. | 12 months post intervention.
  Post-intervention Falls (yes or no)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud Sector III., Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The databases will be available to any interested researcher.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study protocol, Informed Consent Form: available since today. Statistical Analysis Plan: avaliable since may 2024. Clinical Study Report and Analytic Code: avaliable since october 2024.
Access Criteria: Principal investigators of other projects approved by a Clinical Research Ethics Committee will be able to access. They will have access to the previously explained data. The data will be accessible once the project has been published in scientific journals.

REFERENCES:
- [Background] Schoene D, Heller C, Aung YN, Sieber CC, Kemmler W, Freiberger E. A systematic review on the influence of fear of falling on quality of life in older people: is there a role for falls? Clin Interv Aging. 2019 Apr 24;14:701-719. doi: 10.2147/CIA.S197857. eCollection 2019. PMID 31190764
- [Background] Liu TW, Ng GYF, Chung RCK, Ng SSM. Cognitive behavioural therapy for fear of falling and balance among older people: a systematic review and meta-analysis. Age Ageing. 2018 Jul 1;47(4):520-527. doi: 10.1093/ageing/afy010. PMID 29471428
- [Background] Tomita Y, Arima K, Tsujimoto R, Kawashiri SY, Nishimura T, Mizukami S, Okabe T, Tanaka N, Honda Y, Izutsu K, Yamamoto N, Ohmachi I, Kanagae M, Abe Y, Aoyagi K. Prevalence of fear of falling and associated factors among Japanese community-dwelling older adults. Medicine (Baltimore). 2018 Jan;97(4):e9721. doi: 10.1097/MD.0000000000009721. PMID 29369207
- [Background] Makino K, Makizako H, Doi T, Tsutsumimoto K, Hotta R, Nakakubo S, Suzuki T, Shimada H. Impact of fear of falling and fall history on disability incidence among older adults: Prospective cohort study. Int J Geriatr Psychiatry. 2018 Apr;33(4):658-662. doi: 10.1002/gps.4837. Epub 2017 Dec 12. PMID 29231272
- [Background] Lavedan A, Viladrosa M, Jurschik P, Botigue T, Nuin C, Masot O, Lavedan R. Fear of falling in community-dwelling older adults: A cause of falls, a consequence, or both? PLoS One. 2018 Mar 29;13(3):e0194967. doi: 10.1371/journal.pone.0194967. eCollection 2018. PMID 29596521
- [Background] Lee S, Oh E, Hong GS. Comparison of Factors Associated with Fear of Falling between Older Adults with and without a Fall History. Int J Environ Res Public Health. 2018 May 14;15(5):982. doi: 10.3390/ijerph15050982. PMID 29757960
- [Background] Vitorino LM, Teixeira CA, Boas EL, Pereira RL, Santos NO, Rozendo CA. Fear of falling in older adults living at home: associated factors. Rev Esc Enferm USP. 2017 Apr 10;51:e03215. doi: 10.1590/S1980-220X2016223703215. English, Portuguese. PMID 28403369
- [Background] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- [Background] Hughes CC, Kneebone II, Jones F, Brady B. A theoretical and empirical review of psychological factors associated with falls-related psychological concerns in community-dwelling older people. Int Psychogeriatr. 2015 Jul;27(7):1071-87. doi: 10.1017/S1041610214002701. Epub 2015 Jan 30. PMID 25633917
- [Background] Kim JH, Bae SM. Association between Fear of Falling (FOF) and all-cause mortality. Arch Gerontol Geriatr. 2020 May-Jun;88:104017. doi: 10.1016/j.archger.2020.104017. Epub 2020 Jan 27. PMID 32044524
- [Background] Lach HW, Parsons JL. Impact of fear of falling in long term care: an integrative review. J Am Med Dir Assoc. 2013 Aug;14(8):573-7. doi: 10.1016/j.jamda.2013.02.019. Epub 2013 Apr 16. PMID 23602257
- [Background] Alarcon T, Gonzalez-Montalvo JI, Otero Puime A. [Assessing patients with fear of falling. Does the method use change the results? A systematic review]. Aten Primaria. 2009 May;41(5):262-8. doi: 10.1016/j.aprim.2008.09.019. Spanish. PMID 19464526
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Background] Kempen GI, Yardley L, van Haastregt JC, Zijlstra GA, Beyer N, Hauer K, Todd C. The Short FES-I: a shortened version of the falls efficacy scale-international to assess fear of falling. Age Ageing. 2008 Jan;37(1):45-50. doi: 10.1093/ageing/afm157. Epub 2007 Nov 20. PMID 18032400
- [Background] Lee J, Choi M, Kim CO. Falls, a fear of falling and related factors in older adults with complex chronic disease. J Clin Nurs. 2017 Dec;26(23-24):4964-4972. doi: 10.1111/jocn.13995. Epub 2017 Oct 2. PMID 28793363
- [Background] Alcolea-Ruiz N, Alcolea-Ruiz S, Esteban-Paredes F, Beamud-Lagos M, Villar-Espejo MT, Perez-Rivas FJ. [Prevalence of fear of falling and related factors in community-dwelling older people]. Aten Primaria. 2021 Feb;53(2):101962. doi: 10.1016/j.aprim.2020.11.003. Epub 2021 Jan 11. Spanish. PMID 33446358
- [Background] Simsek H, Erkoyun E, Akoz A, Ergor A, Ucku R. Falls, fear of falling and related factors in community-dwelling individuals aged 80 and over in Turkey. Australas J Ageing. 2020 Mar;39(1):e16-e23. doi: 10.1111/ajag.12673. Epub 2019 May 27. PMID 31134742
- [Background] Chang HT, Chen HC, Chou P. Factors Associated with Fear of Falling among Community-Dwelling Older Adults in the Shih-Pai Study in Taiwan. PLoS One. 2016 Mar 2;11(3):e0150612. doi: 10.1371/journal.pone.0150612. eCollection 2016. PMID 26933882
- [Background] Liu JY. Fear of falling in robust community-dwelling older people: results of a cross-sectional study. J Clin Nurs. 2015 Feb;24(3-4):393-405. doi: 10.1111/jocn.12613. Epub 2014 May 2. PMID 24787119
- [Background] Parry SW, Bamford C, Deary V, Finch TL, Gray J, MacDonald C, McMeekin P, Sabin NJ, Steen IN, Whitney SL, McColl EM. Cognitive-behavioural therapy-based intervention to reduce fear of falling in older people: therapy development and randomised controlled trial - the Strategies for Increasing Independence, Confidence and Energy (STRIDE) study. Health Technol Assess. 2016 Jul;20(56):1-206. doi: 10.3310/hta20560. PMID 27480813
- [Background] Zijlstra GA, van Haastregt JC, Ambergen T, van Rossum E, van Eijk JT, Tennstedt SL, Kempen GI. Effects of a multicomponent cognitive behavioral group intervention on fear of falling and activity avoidance in community-dwelling older adults: results of a randomized controlled trial. J Am Geriatr Soc. 2009 Nov;57(11):2020-8. doi: 10.1111/j.1532-5415.2009.02489.x. Epub 2009 Sep 28. PMID 19793161
- [Background] Chua CHM, Jiang Y, Lim S, Wu VX, Wang W. Effectiveness of cognitive behaviour therapy-based multicomponent interventions on fear of falling among community-dwelling older adults: A systematic review and meta-analysis. J Adv Nurs. 2019 Dec;75(12):3299-3315. doi: 10.1111/jan.14150. Epub 2019 Aug 27. PMID 31287182
- [Background] Kruisbrink M, Delbaere K, Kempen GIJM, Crutzen R, Ambergen T, Cheung KL, Kendrick D, Iliffe S, Zijlstra GAR. Intervention Characteristics Associated With a Reduction in Fear of Falling Among Community-Dwelling Older People: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Gerontologist. 2021 Aug 13;61(6):e269-e282. doi: 10.1093/geront/gnaa021. PMID 32267498
- [Background] Duenas EP, Ramirez LP, Ponce E, Curcio CL. [Effect on fear of falling and functionality of three intervention programs. A randomised clinical trial]. Rev Esp Geriatr Gerontol. 2019 Mar-Apr;54(2):68-74. doi: 10.1016/j.regg.2018.09.013. Epub 2018 Nov 24. Spanish. PMID 30482460
- [Derived] Alcolea-Ruiz N, Lopez-Lopez C, Perez-Perez T, Alcolea S, Fearfall Care Clinical Care Group, Perez-Rivas FJ. Effect of a Health Education Intervention to Reduce Fear of Falling and Falls in Older People: A Cluster Randomized Clinical Trial Protocol. Healthcare (Basel). 2024 Dec 11;12(24):2510. doi: 10.3390/healthcare12242510. PMID 39765937
- See also: Preocupación a caer validación de un instrumento de medición en personas mayores chilenas que viven en la comunidad — https://dialnet.unirioja.es/servlet/articulo?codigo=6185112